CLINICAL TRIAL: NCT03412500
Title: A Comparative Efficacy Study of Vancomycin Dosage Adjustment by Equation-based Method and Vancomycin Trough Concentration Method for Treatment of Infections Caused by Methicillin Resistant Staphylococcus Aureus
Brief Title: Vancomycin Dosage Adjustment for MRSA Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pinyo Rattanaumpawan (Other)
Responsible Party: Sponsor-Investigator, Pinyo Rattanaumpawan, Assistant Professor, Siriraj Hospital
Organization: Siriraj Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101/2559(EC1)
Record Dates: First submitted 2016-06-03; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: Methicillin-Resistant Staphylococcus aureus; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin trough concentration method (Active Comparator): vancomycin dosage will be adjusted by the trough concentration method
  Interventions: Drug: Vancomycin trough concentration method
- Vancomycin equation-based method (Experimental): vancomycin dosage will be adjusted by the equation-based method
  Interventions: Drug: Vancomycin equation-based method

INTERVENTIONS:
Drug: Vancomycin equation-based method — Vancomycin dosage will be adjusted according to the equation-based method
  Other Names: intervention arm
  Arms: Vancomycin equation-based method
Drug: Vancomycin trough concentration method — Vancomycin dosage will be adjusted according to the trough concentration method
  Other Names: control arm
  Arms: Vancomycin trough concentration method

SUMMARY:
An open-label randomized controlled trial to compare two vancomycin dosage adjustment methods

DETAILED DESCRIPTION:
An open-label randomized controlled trial to compare two vancomycin dosage adjustment methods; a vancomycin trough concentration method and a equation-based method.

ELIGIBILITY:
Inclusion Criteria:

1. Thai hospitalized patients, age>18 years
2. Require vancomycin therapy ≥ 3 days
3. Documented MRSA infection including pneumonia, bacteremia, intra-abdominal infection or skin and soft tissue infection
4. Have been checked for serum creatinine within 48 hours and serum albumin within 7 days prior to enrollment
5. Received an appropriate loading dose of vancomycin
6. Have been treated with an appropriate maintenance dose of vancomycin
7. Willing to sign an informed consent

Exclusion Criteria:

1. CrCl< 10 ml/min or receiving renal replacement therapy
2. Pregnancy or lactation
3. Actual BW> 90 kg
4. Serum albumin <2 g/dl
5. Having an active cancer or receiving chemotherapy
6. Hx of vancomycin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Clinical response | End of therapy (an average of 2 weeks)
  Clinical response will be evaluated at the end of therapy (EOT) by a clinician investigator. Clinical response will be classified as good clinical response, partial clinical response, poor clinical response and undetermined.

SECONDARY OUTCOMES:
Renal adverse event | Day 5 after vancomycin therapy
  Double serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: pinyo rattanaumpawan, md, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No